CLINICAL TRIAL: NCT05344690
Title: Evaluation of the Relationship Between SLMAP and EPO Genetic Polymorphism and the Risk of Diabetic Retinopathy in Egyptian Diabetic Patients: A Case-Control Study
Brief Title: SLMAP and EPO Genetic Polymorphism in Diabetic Retinopathy
Status: Completed | Type: Observational
Sponsor: Ain Shams University (Other)
Responsible Party: Principal Investigator, Rana Sayed Fouad, Principal investigator, Ain Shams University
Other Study IDs: RHDIRB2020110301 REC 72
Record Dates: First submitted 2022-04-19; First posted 2022-04-25 (Actual); Last update posted 2024-02-07 (Actual); Status verified 2024-02

CONDITIONS: Diabetic Retinopathy
MeSH Terms: conditions — Diabetic Retinopathy

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- cases: diabetic patients suffering from clinically confirmed diabetic retinopathy
  Interventions: Genetic: SLMAP and EPO genetic polymorphism
- controls: matched (based on gender and duration of diabetes) diabetic patients free from diabetic retinopathy will be recruited.
  Interventions: Genetic: SLMAP and EPO genetic polymorphism

INTERVENTIONS:
Genetic: SLMAP and EPO genetic polymorphism — Presence of EPO gene SNP rs551238 and SLMAP rs17058639 gene polymorphisms

SUMMARY:
A case-control study to assess the association between the risk of diabetic retinopathy in Egyptians and genetic polymorphism of both EPO and SLMAP genes.

DETAILED DESCRIPTION:
Traditional environmental risk factors, such as glycemic control and duration of diabetes, failed to fully explain why some individuals remain protected while others progress to severe diabetic retinopathy.

Several studies suggest variations in diabetic retinopathy prevalence depending on racial background and genetic polymorphism.

ELIGIBILITY:
Inclusion Criteria:

* Age >30-60
* Type 2 DM
* Duration of diabetes from 5-10 years
* Egyptian patients

Exclusion Criteria:

* Other ophthalmic diseases not related to diabetes

Ages: 30 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: All diabetic patients registered to the outpatient clinic of the Endocrinology Unit will be assessed for eligibility followed by screening for diabetic retinopathy by fundoscopic examination Those with diabetic retinopathy will be assigned to the case group while matched diabetic patients free from diabetic retinopathy will be assigned to the control group.
Sampling Method: Non-Probability Sample
Enrollment: 180 (Actual)
Dates: Start 2022-05-20 (Actual); Primary Completion 2023-04-30 (Actual); Study Completion 2023-06-30 (Actual)

PRIMARY OUTCOMES:
Association of SLMAP gene polymorphism and the risk of confirmed diabetic retinopathy diagnosis | At baseline (upon confirmed diagnosis of diabetic retinopathy)
  the odds ratio of being diagnosed with diabetic retinopathy in those with SLMAP rs17058639 single nucleotide polymorphism compared to wild type
Association of EPO gene polymorphism and the risk of confirmed diabetic retinopathy diagnosis | At baseline (upon confirmed diagnosis of diabetic retinopathy)
  The odds ratio of being diagnosed with diabetic retinopathy in those with EPO rs551238 single nucleotide polymorphism compared to wild type

SECONDARY OUTCOMES:
The association of confounding factors on the incidence of diabetic retinopathy | At baseline
  A multiple logistic regression model will be fitted to assess the association of diabetic retinopathy to confounders (microalbuminuria, lipid profile, age, gender,...etc.)

CONTACTS AND LOCATIONS:
Overall Officials: Lamiaa M El Wakeel, PhD, Study Chair — Faculty of Pharmacy, Ain Shams University
Locations (1):
- Ain Shams University Hospitals, Cairo, Abbasseya, Egypt

IPD SHARING:
Plan to Share IPD: Undecided